CLINICAL TRIAL: NCT04792385
Title: A Multicenter, Open-label, Single-Arm Study to Evaluate the Safety, Compliance and Pharmacokinetics Associated With the Use of a Combined Oral Contraceptive Containing 15 mg Estetrol Monohydrate and 3 mg Drospirenone in Post-menarchal Female Adolescents for 6 Cycles
Brief Title: Safety, Compliance and Pharmacokinetics of Estetrol Monohydrate/Drospirenone 15/3 mg in Post-menarchal Female Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Estetra (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MIT-Es001-C303; 2019-003002-27 (EudraCT Number)
Record Dates: First submitted 2021-03-05; First posted 2021-03-11 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Safety
Keywords: Estetrol; Drospirenone; Combined oral contraceptive; Oral contraception; Cycle control; Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- E4/DRSP 15/3 mg (Experimental): Single treatment arm will receive E4/DRSP 15/3 mg
  Interventions: Drug: E4/DRSP 15/3 mg combined tablet

INTERVENTIONS:
Drug: E4/DRSP 15/3 mg combined tablet — One E4/DRSP 15/3 mg combined tablet once per day for 24 days followed by 4 days of placebo tablets; this 28-day cyclic regimen should be taken for 6 consecutive cycles.
  Other Names: 15 mg estetrol monohydrate/3 mg drospirenone combined oral contraceptive

SUMMARY:
To evaluate the safety, compliance, and pharmacokinetics profile of estetrol monohydrate (E4) 15 mg combined with drospirenone (DRSP) 3 mg in post-menarchal participants between the age of 12 and 17 years + 2 months.

DETAILED DESCRIPTION:
This is a Phase 3, open-label, non-controlled study in healthy post-menarchal female participants who will be enrolled to receive once daily E4/DRSP 15/3 mg for six (6) 28-day cycles in a 24/4-day regimen (i.e. 24 days of active tablets followed by 4 days of placebo tablets [4-day hormone-free interval]). The study will include 6 visits:

At screening visit (Visit 1), informed consent will be signed by the participants and their parent(s) or legal representative(s) and the screening procedures will be performed. The site will also complete an Eligibility confirmation phone call to the participant after Visit 1. During the enrollment visit (Visit 2, between Days 12 and 19 of the pre-treatment cycle), eligibility criteria will be reviewed and the participant participation will be confirmed. Participants will be trained in the use of an electronic diary and will receive the study drug. A follow-up call will be performed after Visit 2, within 7 days following the first investigational product intake. Afterwards, the participants will attend 3 on-treatment visits at the clinical site [between Days 14 and 21 of the Cycle 1(Visit 3), Cycle 3 (Visit 4), and Cycle 6 (Visit 5)] and one visit after end of Cycle 6 (Visit 6).

For participants who consent to participate in a pharmacokinetics sub-study, blood samples for this sub-study will be taken at Visit 3 and Visit 5.

Adverse events will be followed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Post-menarchal female participant requesting combined oral contraceptive (COC) either for contraceptive or for therapeutic use.
2. Negative serum pregnancy test at screening and negative urine pregnancy test at enrollment.
3. Aged 12 to 17 years and 2 months (inclusive) [Estonia-specific: 15 to 17 years and 2 months (inclusive)] at the time of signing the informed consent.
4. Willing to use the investigational product for 6 consecutive cycles.
5. Good physical and mental health on the basis of medical, surgical and gynecological history, physical examination, clinical laboratory, and vital signs.
6. Body mass index (BMI) below or equal to the percentile 97 (P97) on the local pediatric BMI curves.
7. Able to fulfill the requirements of the protocol, undergo all study procedures including e-diary and questionnaires completion.
8. Having indicated the willingness to participate in the study by providing written assent.
9. Having parent(s) or legal representative(s) willing and able to provide written informed consent.

Exclusion Criteria:

1. For participants who are not using hormonal contraception at screening, a menstrual cycle length shorter than 21 days or longer than 45 days.
2. Currently using an injectable or a dermally implantable hormonal method of contraception.
3. Known hypersensitivity to any of the investigational product ingredients.
4. Currently pregnant or breastfeeding or with the intention to become pregnant during the course of the study.
5. Less than 6 weeks since last delivery/2nd trimester abortion and before spontaneous menstruation has occurred following a delivery or 2nd trimester abortion.
6. Any condition representing a contraindication / precaution to the use of COCs, including but not limited to:

   1. dyslipoproteinaemia,
   2. diabetes mellitus with vascular involvement (nephropathy, retinopathy, neuropathy, other),
   3. arterial hypertension (controlled and uncontrolled)
   4. personal or first-degree family history of deep vein thrombosis or pulmonary embolism,
   5. current or planned prolonged immobilization,
   6. known inherited or acquired hypercoagulopathies or thrombogenic mutations (e.g. Factor V Leiden mutation),
   7. current treatment with anticoagulants,
   8. presence or history of arterial thromboembolism,
   9. complicated valvular heart disease,
   10. systemic lupus erythematosus,
   11. presence or history of migraine with aura,
   12. symptomatic gallbladder disease,
   13. porphyria.
7. Within the past 6 months, undiagnosed (unexplained) abnormal vaginal bleeding, or any abnormal bleeding that could possibly recur during the study.
8. Presence or history of recurrent pelvic inflammatory disease.
9. Any clinically relevant lower genital tract infection (including gonorrhea and chlamydia infections) until successfully treated, in the opinion of the Investigator.
10. Presence or history of hepatic disease as long as liver function values have not returned to normal.
11. Renal impairment
12. Hyperkalemia or presence of conditions that predispose to hyperkalemia such as renal impairment, hepatic impairment, adrenal insufficiency and daily, long-term treatment for chronic conditions or diseases with medications that may increase serum potassium concentration (e.g. angiotensin-converting-enzyme (ACE) inhibitors, angiotensin-II receptor antagonists, potassium-sparing diuretics, potassium supplementation, heparin, aldosterone antagonist and non-steroidal anti-inflammatory drugs).
13. History of organ transplantation within 5 years before screening or chronic disease potentially necessitating organ transplantation during the anticipated course of the study.
14. Presence or history of sex hormone-related malignancy.
15. History of non-hormone-related malignancy within 5 years before screening.
16. Current regular use or regular use within 1 month prior to Visit 2 of drugs potentially triggering interactions with COCs including but not limited to:

    1. Cytochrome P450 3A4 (CYP 3A4) inducers: barbiturates, primidone, bosentan, felbamate, griseofulvin, oxcarbazepine, topiramate, carbamazepine, phenytoin, rifampicin, St John's wort (Hypericum perforatum L).
    2. CYP 3A4 inhibitors: azole antifungals excluding topical fluconazole, phenylbutazone, modafinil, cimetidine, verapamil, macrolides excluding azithromycin, diltiazem and grapefruit juice.
    3. Human immunodeficiency virus (HIV)/Hepatitis C virus (HCV) protease inhibitors and non-nucleoside reverse transcriptase inhibitors.
17. History of alcohol or drug abuse (including laxatives) within 12 months prior to screening.
18. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs.
19. Uncontrolled thyroid disorders.
20. Participation in another investigational drug clinical study within 1 month (30 days) or have received an investigational drug within the last month (30 days) prior to screening.
21. Sponsor, Contract Research Organization (CRO) or Investigator's site personnel directly affiliated with this study.
22. The participant is judged by the Investigator to be unsuitable for any reason.
23. [Estonia-specific: Subjects who are at a gynecologist visit for the first time in their life may not sign the informed consent during this first visit.]

Ages: 12 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 145 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2023-11-24 (Actual); Study Completion 2023-11-24 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events | From Cycle 1 to end of study (between Days 16 and 23 of Cycle 7) (each cycle is 28 days)
  Treatment emergent adverse events (TEAEs) are those adverse events occurring from time point of first ingestion of the investigational product until last visit or any event already present that worsens in either intensity or frequency following exposure to the treatment.
Number of participants with treatment-emergent adverse events related to the investigational product | From Cycle 1 to end of study (between Days 16 and 23 of Cycle 7) (each cycle is 28 days)
  Treatment emergent adverse events (TEAEs) are those adverse events occurring from time point of first ingestion of the investigational product until last visit or any event already present that worsens in either intensity or frequency following exposure to the treatment.
  The causality of TEAEs (related or not related) is based on the following considerations: associative connections (time and/or place), pharmacological explanations, previous knowledge of the drug, presence of characteristic clinical or pathological phenomena, exclusion of other causes, and/or absence of alternative explanations.
Number of participants with abnormal physical examination results | At Baseline and at the end of treatment (Cycle 6) (each cycle is 28 days)
  The physical examination will include an evaluation of the following: body as a whole, skin, head, eyes, ears, nose, and throat, neck, cardiovascular, respiratory, musculoskeletal, neurologic, lymphatic/thyroid, abdomen.
Number of participants with abnormal vital sign results | From Baseline to end of treatment (Cycle 6) (each cycle is 28 days)
  Vital signs will include sitting systolic and diastolic blood pressures and heart rate.
Number of participants with abnormal electrocardiogram (ECG) results | At Baseline and at the end of treatment (Cycle 6) (each cycle is 28 days)
  The ECG interpretation scheme will include the analysis of the morphology, rhythm, conduction, ST segment, PR, QRS, QT and QTc (according to QTcFrid) intervals, T waves, U waves and the presence or absence of any pathological changes.
Number of participants with abnormal clinical laboratory assessment results | At Baseline and at the end of treatment (Cycle 6) (each cycle is 28 days)
  Laboratory assessment will include blood hematology and biochemistry.

SECONDARY OUTCOMES:
Percentage of compliance by cycle [Estonia-specific: and overall compliance] | At Cycles 1, 2, 3, 4, 5 ,6 (each cycle is 28 days)
  The percentage of compliance per cycle is calculated as the ratio of the total number pills taken during the cycle based on the daily response values entered by the participant in the e-diary and the number of pills expected to be taken during the cycle based on the total number of treatment days.
  [Estonia-specific: the percentage of overall compliance is calculated as the ratio of the total number of pills taken across all cycles based on the daily response values entered by the participant in the e-diary and the number of pills expected to be taken from the start date of cycle 1 until the day of the last dose.]
Mean plasma estetrol (E4) concentration | At Cycle 1 and at the end of treatment (Cycle 6) (each cycle is 28 days)
Mean plasma drospirenone (DRSP) concentration | At Cycle 1 and at the end of treatment (Cycle 6) (each cycle is 28 days)
Number of participants with unscheduled bleeding and/or spotting episodes | At Cycles 1,2, 3, 4, 5, 6 (each cycle is 28 days)
Number of participants with absence of bleeding/spotting episodes | At Cycles 1,2, 3, 4, 5, 6 (each cycle is 28 days)
Mean number of unscheduled bleeding and spotting days per cycle | At Cycles 1,2, 3, 4, 5, 6 (each cycle is 28 days)
Mean number of scheduled bleeding and spotting days per cycle | At Cycles 1,2, 3, 4, 5, 6 (each cycle is 28 days)
Change in the Score of the Menstrual Distress Questionnaire (MDQ) from baseline to Cycles 1, 3 and 6 | At Baseline and at Cycles 1, 3 and 6 (each cycle is 28 days)
  The MDQ is a standard method for measuring cyclical perimenstrual symptoms. The participants will rate common symptoms and feelings associated with menstruation using the following scale: 0 (no experience of symptom), 1 (present, mild), 2 (present, moderate), 3 (present, strong),and 4 (present, severe) observed during pre-menstrual (4 days before menstruation), menstrual (most recent flow) and intermenstrual (remainder of the cycle) phases.
Change in the Visual Analogue Scale (VAS) score of dysmenorrhea from baseline to Cycles 1, 3 and 6 | At Baseline, Cycles 1, 3, and at the end of treatment (Cycle 6) (each cycle is 28 days)
  Each day participants will be asked to score their menstruation pain of the previous 24 hours using a scale from 0 to 10, with 0 = no hurt and 10 = hurts worst.
Change in the number of days with dysmenorrhea from baseline to Cycles 1, 3 and 6 | At Baseline, Cycles 1, 3, and at the end of treatment (Cycle 6) (each cycle is 28 days)
Number of participants who will use rescue medication for dysmenorrheal pain from baseline to Cycles 1, 3 and 6 | At Baseline, Cycles 1, 3, and at the end of treatment (Cycle 6) (each cycle is 28 days)
Change in Health Questionnaire for children and Young People (KIDSCREEN-27 questionnaire) from baseline to Cycles 1, 3 and 6 | At Baseline, Cycles 1, 3, and at the end of treatment (Cycle 6) (each cycle is 28 days)
  KIDSCREEN-27 is a validated health-related quality of life questionnaire developed for children and adolescents. This questionnaire measures five Rasch scaled dimensions of well-being including: (1) Physical Well-being (5 items), (2) Psychological Well-being (7 items), (3) Autonomy and Parents (7 items), (4) Peers and Social Support (4 items), and (5) School Environment (4 items). Responses are indicated using a 5-point ordinal scale with responses ranging from 'never' to 'always', 'not at all' to 'extremely', or 'poor' to 'excellent'.
Change in sex-hormone binding globulin (SHBG) level from baseline to Cycle 6 | At Baseline and at the end of treatment (Cycle 6) (each cycle is 28 days)
Change in Activated protein C resistance endogenous thrombin potential based (APCr [ETP based]) level from baseline to Cycle 6 | At Baseline and at the end of treatment (Cycle 6) (each cycle is 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Estetra, Study Director — Estetra
Locations (21):
- Estonia (4):
  - KVL Medical Office/KVL Arstikabinet, Pärnu
  - East-Tallinn Central Hospital, Tallinn
  - Sexual Health Clinic, Tallinn, Tallinn
  - Sexual Health Clinic, Tartu, Tartu
- Finland (3):
  - VL-Medi Oy, Helsinki
  - Lääkärikeskus Mehiläinen, Kuopio
  - Lääkärikeskus Gyneko, Oulu
- Georgia (2):
  - Estetra Study Site, Batumi
  - Estetra Study Site, Tbilisi
- Latvia (2):
  - A. Krumpane practice, Daugavpils
  - Childrens Clinical University Hospital, Riga
- Poland (7):
  - Estetra Study Site, Bialystok
  - Estetra Study Site, Katowice
  - Estetra Study Site, Lublin
  - Estetra Study Site, Ostrowiec Świętokrzyski
  - Estetra Study Site, Poznan
  - Estetra Study Site, Raszyn
  - Estetra Study Site, Wroclaw
- Sweden (3):
  - Akardo Medsite at Sturebadet Health Care, Stockholm
  - Karolinska University, Department of Gynecology and Reproductive Medicine, Stockholm
  - Karolinska University, WHO Center, Stockholm